CLINICAL TRIAL: NCT02852330
Title: Intracochlear Potentials: Intraoperative and Post-operative Measurement Clinical Investigation
Brief Title: Intracochlear Potentials: Volta Study
Acronym: CLTD5663
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: The Hearing Cooperative Research Centre (Other); Royal Victoria Eye and Ear Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CLTD5663; CLTD5663 (Other: Cochlear)
Record Dates: First submitted 2016-06-03; First posted 2016-08-02 (Estimated); Results first posted 2021-05-25 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2022-10

CONDITIONS: Hearing Loss
Keywords: Voltage tomography
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Voltage tomography (Experimental): Voltage tomography measurements will be made with the SA16 research software and CS19 (1.6.2) software during and/or immediately after electrode insertion during cochlear implantation and at scheduled post-operative clinical visits.
  Interventions: Device: SA16 research software; Device: CS19 (1.6.2)

INTERVENTIONS:
Device: SA16 research software — Software for measurement of voltage tomography intraoperatively.
Device: CS19 (1.6.2) — Software for measurement of voltage tomography post-operatively.

SUMMARY:
Collection of normative voltage tomography data during and/or immediately after electrode insertion into the cochlea using Surgical Assistant (SA16) research software and postoperatively at activation, three and twelve months post-activation with CS19 research software in adults who are receiving a Cochlear Nucleus CI512, CI422, CI522 or CI532 cochlear implant.

DETAILED DESCRIPTION:
The clinical investigation will gather impedance and transimpedance (voltage tomography) data intraoperatively and post-operatively which can be used to characterize the electrical properties of the living cochlea.

The Surgical Assistant Research Tool (SA16) research software is a software tool developed by Cochlear Limited. The use of the SA16 research software in the current clinical investigation is intended to support Cochlear's research into the development of implant telemetry based surgical tools.

The SA16 research software is designed to perform a series of predefined measurements with minimal intervention both during and immediately following electrode insertion using telemetry from the implant via the Sound Processor to the computer. These measurements include real time continuous measurements, intended for use during the electrode insertion portion of the surgical procedure, and baseline measurements following the completion of electrode insertion.

The SA16 research software will be used in the current clinical investigation in adults who meet current indications for cochlear implantation in Australia. The SA16 research software is not for use with patients who are receiving an implant that directly contacts neural tissue, such as auditory brainstem implants (ABI).

CS19 (1.6.2) software will be used to collect voltage tomography measurements post-implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Meet current cochlear implant indications at the implanting centre for a Cochlear Nucleus CI512, CI422, CI522 or CI532 cochlear implant
2. Aged 18 years and older at the time of implantation.

Exclusion Criteria:

1. Recipient of a Nucleus 24 ABI device
2. Medical or psychological conditions that contraindicate undergoing general anaesthesia or surgery.
3. Ossification, malformation or any other cochlear anomaly, such as common cavity, that might prevent complete insertion of the electrode array, as confirmed by medical examination.
4. Unwillingness or inability of the candidate to comply with all investigational requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cowan, Principal Investigator — The HEARing CRC; Robert Briggs, Principal Investigator — The Royal Victorian Eye and Ear Hospital
Locations (2):
- Australia (2):
  - The Hearing Cooperative Research Centre, Carlton, Victoria
  - Royal Victorian Eye and Ear Hospital, East Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Voltage Tomography
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Voltage Tomography
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 70.3 [50 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 20

OUTCOME MEASURES:

1. Primary Outcome: Normative Voltage Tomography Data
Description: Gather normative voltage tomography data for retrospective analysis. After insertion of the electrode array, TIM measurements will be taken from each subject using the cochlear implant system and Surgical Assistant Research Tool software. A Tip Foldover (TFO) in the software and x-rays will be used to identify any occurrence of a tip foldover.
Time Frame: intraoperatively during and/or immediately after electrode insertion into the cochlea, with a measurement time of approximately 10 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Voltage Tomography
Number analyzed (Participants) | 20
Participants
  Nominal TIMs | 19
  Anomalous TIMs | 1
  Correct TIP detection | 19
  Incorrect TIP detection | 1

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Voltage Tomography
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voltage Tomography (N=20)
Cardiac arrest (Cardiac disorders) | 1 (1) — Cardiac arrest during hip replacement surgery, resulting in cochlear implant surgery cancellation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT02852330/Prot_002.pdf